CLINICAL TRIAL: NCT00167752
Title: Quality of Life, Emotional and Sleep Problems in Chronic Skin Diseases
Brief Title: Psychiatric Problems in Chronic Skin Diseases
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2002-0420
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Psoriasis; Acne; Vitiligo; Atopic Dermatitis; Pruritic Dermatitis
MeSH Terms: conditions — Psoriasis; Acne Vulgaris; Vitiligo; Dermatitis, Atopic; Pruritus

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to investigate the prevalence of depression, anxiety, and sleep problems in patients with chronic skin diseases in dermatology clinics at the University of Wisconsin Hospital and Clinics.

ELIGIBILITY:
Inclusion Criteria:

* Subjects suffering from a chronic skin condition that has lasted over six months

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-12; Primary Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ladan Mostaghimi, MD, Principal Investigator — University of Wisconsin, Madison